CLINICAL TRIAL: NCT04156724
Title: Helmet Ventilation During Self-Paced Walking Test With Chronic Obstructive Pulmonary Disease
Brief Title: Helmet Ventilation During Self-Paced Walking Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Leader of Respiratory Therapist, Fu Jen Catholic University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: C108032
Record Dates: First submitted 2019-11-06; First posted 2019-11-07 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HV (Experimental): 6MWT with helmet ventilation
  Interventions: Device: Helmet vetilation
- Control (No Intervention): 6MWT alone according to ATS guideline

INTERVENTIONS:
Device: Helmet vetilation — We will apply non-invasive positive pressure ventilation via a helmet as interface
  Arms: HV

SUMMARY:
The aim of this study is to investigate the use helmet ventilation (HV) in walking test and analysis of effect patients with COPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is characterized by persistent airflow limitation with chronic inflammation of the respiratory system. Symptoms of COPD may contribute to activity restriction, deconditioning and exercise intolerance. Non-invasive positive pressure ventilation (NIPPV) has been shown to improve exercise intolerance and health-related quality of life in patients with severe COPD. Helmet ventilation (HV) is a new option for NIPPV to alternative to nasal or face mask. A study which published on JAMA demonstrated the feasibility and benefits of HV. The aim of this study is to investigate the use helmet ventilation (HV) in walking test and analysis of effect patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Patents with COPD who confirm by pulmonary function test

Exclusion Criteria:

* COPD AE within 3 months
* Diagnosed neuromuscular disease
* Unable to perform 6-MWT

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
6WMD | 2 days
  Walking distance of six minute walking test

SECONDARY OUTCOMES:
Heart rate | 2 days
  Heart rate of six minute walking test
Respiratory rate | 2 days
  Respiratory rate of six minute walking test
modified Borg dyspnea scale | 2 days
  A self report level of dyspnea score ranging from 0 to 10, 0 represent no dyspnea and 10 represents the worse

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Lun Liu, MD, Principal Investigator — Department of Emergency and Critical Care Medicine, Fu Jen Catholic University Hospital
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel BK, Wolfe KS, Pohlman AS, Hall JB, Kress JP. Effect of Noninvasive Ventilation Delivered by Helmet vs Face Mask on the Rate of Endotracheal Intubation in Patients With Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. JAMA. 2016 Jun 14;315(22):2435-41. doi: 10.1001/jama.2016.6338. PMID 27179847
- [Background] Patel BK, Wolfe KS, MacKenzie EL, Salem D, Esbrook CL, Pawlik AJ, Stulberg M, Kemple C, Teele M, Zeleny E, Macleod J, Pohlman AS, Hall JB, Kress JP. One-Year Outcomes in Patients With Acute Respiratory Distress Syndrome Enrolled in a Randomized Clinical Trial of Helmet Versus Facemask Noninvasive Ventilation. Crit Care Med. 2018 Jul;46(7):1078-1084. doi: 10.1097/CCM.0000000000003124. PMID 29595563
- [Background] Dreher M, Storre JH, Windisch W. Noninvasive ventilation during walking in patients with severe COPD: a randomised cross-over trial. Eur Respir J. 2007 May;29(5):930-6. doi: 10.1183/09031936.00075806. Epub 2007 Mar 1. PMID 17331969
- [Derived] Chao KY, Liu WL, Nassef Y, Lai PZ, Wang JS. A pilot crossover trial assessing the exercise performance patients chronic obstructive pulmonary disease. Sci Rep. 2022 Mar 9;12(1):4158. doi: 10.1038/s41598-022-07698-z. PMID 35264615